CLINICAL TRIAL: NCT01293760
Title: Immediate Post-placental Insertion of the Copper T 380A After Cesarean Delivery Versus 6 Week Post-cesarean Insertion: A Pilot Randomized Controlled Trial
Brief Title: Immediate Post-placental Insertion of the Copper T 380A After Cesarean Delivery Versus 6 Week Post-cesarean Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planned Parenthood League of Massachusetts (Other)
Collaborators: Mulago Hospital, Uganda (Other); Brigham and Women's Hospital (Other); Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2010p001355
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Contraception
Keywords: intrauterine device; contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6 weeks interval insertion (Other): IUD is inserted 6 weeks following c-section delivery of baby and placenta
  Interventions: Other: 6 weeks interval insertion
- Immediate insertion (Experimental): IUD is inserted immediately following c-section delivery of baby and placenta
  Interventions: Other: Immediate insertion

INTERVENTIONS:
Other: Immediate insertion — Insertion of Copper T 380A immediately after c-section delivery of baby and placenta
  Arms: Immediate insertion
Other: 6 weeks interval insertion — Insertion of Copper T 380A 6 weeks after c-section delivery of baby and placenta
  Arms: 6 weeks interval insertion

SUMMARY:
The purpose of this study is to determine, in a pilot setting, if this study is feasible in terms of recruitment, willingness to be randomized, provision of contraceptive methods, and follow-up. The investigators hypothesize that this pilot study will be feasible in terms of recruitment, provision of care, and follow-up.

The study will be a pilot randomized controlled trial comparing outcomes of immediate post-placental insertion of the Copper T 380A (Group 1) to outcomes of interval insertion of the Copper T 380A performed 6 weeks after delivery (Group 2) for patients undergoing scheduled cesarean delivery at Mulago Hospital in Kampala, Uganda. This study will not be powered to detect a difference, but rather the investigators will enroll all eligible and interested women during the three-month enrollment period. Potential participants who do not choose an IUD or who choose not to participate will be offered an anonymous opt-out survey.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant at time of enrollment
2. Scheduled to undergo non-emergent cesarean delivery
3. Will have to wait at least 8 hours before their cesarean section
4. Are not in active labor
5. Desires to use the Copper T 380A for contraception
6. Willing and able to sign an informed consent
7. Willing to comply with the study protocol
8. Age greater than or equal to 18 years
9. English or Luganda speaking
10. Willing to be accompanied home upon discharge from the hospital and have their address recorded in order to be able to visit them at home at 6 months postpartum if they do not return for their 6 month follow-up visit.

Exclusion Criteria:

1. Allergy to copper or pelvic tuberculosis, severe thrombocytopenia
2. Positive N. gonorrheae or C. trachomatis testing
3. Presence of leiomyomata significantly distorting the uterine cavity and thus not allowing placement of the Copper T 380A
4. Uterine anomaly which would not allow placement of the Copper T 380A
5. Current cervical cancer or carcinoma in-situ
6. Desire for repeat pregnancy in less than 12 months
7. Evidence of intra-uterine infection (Chorioamnionitis)
8. Pre-term birth prior to 34 weeks of gestation
9. Diagnosis of AIDS (HIV is not an exclusion criteria)
10. Fetal demise
11. Antepartum hemorrhage
12. Ruptured uterus
13. Eclampsia
14. Evidence of severe anemia

Post enrollment exclusion criteria

1. Group 1: Interval development of any of the above exclusion criteria (New evidence of chorioamnionitis; fetal demise; ruptured uterus; eclampsia; severe anemia)
2. Group 1: Post-partum hemorrhage with continued active bleeding that does not allow placement of the Copper T 380A within 10 minutes of the delivery of the placenta
3. Group 1: Prolonged rupture of membranes > 12 hours
4. Group 2: Diagnosis of active cervical infection within 3 months of planned insertion, or evidence of active pelvic or cervical infection, pus at the cervical os or any concern for upper genital tract infection, including fever (temperature ≥ 38° C) or uterine or adnexal tenderness. Diagnosis of new pregnancy.
5. Group 2: Interval development of any of the above exclusion criteria (i.e. new suspicion of cervical cancer or carcinoma in situ)
6. Both Groups: Participant no longer desires a Copper T 380A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
6 month IUD usage rates | 6 months
  The number of participants enrolled who are using the Copper T 380A at 6 months post-delivery. This will include participants who are excluded at time of delivery or interval insertion and participants who do not follow up for interval Copper T 380A insertion

SECONDARY OUTCOMES:
IUD Expulsion | within 6 months
  The time until expulsion of the Copper T 380A will be defined as the time from insertion until expulsion occurred, if known. If the date of expulsion is not known, this will be documented as the day after the IUD was last known to be in place. If a pregnancy is detected and the Copper T 380A is absent (and the participant was unaware of expulsion), the expulsion will be assumed to have occurred at the time of conception, as determined by gestational age on ultrasound. Expulsions will be measured as total expulsions and separately noted whether complete or partial
IUD Removal | within six months
  The proportion of participants who have the Copper T 380A inserted and who deliberately have it removed. We will also analyze the time to removal for these participants
IUD insertion | within 6 months
  The proportion of participants receiving a Copper T 380A in each group
Pregnancy | within 6 months
  Time to pregnancy will be calculated from the date of delivery until the estimated date of conception of a subsequent pregnancy, as based on sonographic dating. If sonographic dating is not available, the date of the last missed menses or three weeks before the first positive urine pregnancy test (if amenorrheic or oligomenorrheic) will be used
Infection | within 6 months
  The diagnosis of PID will be made based on the 2006 CDC guidelines and the criteria used in the PEACH study
Uterine Perforation | within 6 months
  The diagnosis of a perforation may be made by a transvaginal sonogram that shows no Copper T 380A within the uterus and an abdominal radiograph that shows a Copper T 380A within the abdominal cavity

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Planned Parenthood League of Massachusetts
Locations (1):
- Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Derived] Sothornwit J, Kaewrudee S, Lumbiganon P, Pattanittum P, Averbach SH. Immediate versus delayed postpartum insertion of contraceptive implant and IUD for contraception. Cochrane Database Syst Rev. 2022 Oct 27;10(10):CD011913. doi: 10.1002/14651858.CD011913.pub3. PMID 36302159
- [Derived] Lester F, Kakaire O, Byamugisha J, Averbach S, Fortin J, Maurer R, Goldberg A. Intracesarean insertion of the Copper T380A versus 6 weeks postcesarean: a randomized clinical trial. Contraception. 2015 Mar;91(3):198-203. doi: 10.1016/j.contraception.2014.12.002. Epub 2014 Dec 12. PMID 25499587